CLINICAL TRIAL: NCT06571045
Title: A Randomized, Double-Masked, Multi-Center, 3-Arm Pivotal Phase 2/3 Study to Evaluate The Efficacy and Safety of Intravitreal EYE103 Compared With Intravitreal Ranibizumab (0.5mg) in Participants With Diabetic Macular Edema
Brief Title: A Study to Evaluate the Efficacy and Safety of 2 Doses of EYE103 Compared With Ranibizumab (0.5 mg) in Participants With DME
Acronym: BRUNELLO
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: EyeBiotech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EYE-RES-102
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Macular Edema (DME)
Keywords: Diabetic Macular Edema; DME
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Intervention Model Description: Parallel enrollment into 1 of 3 arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- EYE103 Low Dose Treatment Arm (Experimental): EYE103 Low Dose Treatment Arm
  Interventions: Drug: EYE103
- EYE103 High Dose Treatment Arm (Experimental): EYE103 High Dose Treatment Arm
  Interventions: Drug: EYE103
- Ranibizumab Treatment Arm (Active Comparator): Ranibizumab Treatment Arm
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab is a commercially available anti-VEGF treatment formulated for intravitreal administration for use in patients with diabetic macular edema
  Other Names: Lucentis
  Arms: Ranibizumab Treatment Arm
Drug: EYE103 — EYE103 is a humanized antibody formulated for intravitreal administration
  Other Names: Restoret
  Arms: EYE103 High Dose Treatment Arm; EYE103 Low Dose Treatment Arm

SUMMARY:
EYE-RES-102 is a randomized, double masked pivotal study to evaluate the efficacy and safety of 2 dose levels of EYE103 in comparison with the active control, ranibizumab, in patients with diabetic macular edema (DME)

In the first year, all 3 treatment groups will be treated every 4 weeks with either EYE103 or ranibizumab. Beginning at Year 2, the frequency of treatment for participants will shift based on a personalized treatment interval algorithm.

Approximately 960 participants will be entered in the study.

DETAILED DESCRIPTION:
EYE-RES-102 is a randomized, double masked pivotal study to evaluate the efficacy and safety of 2 dose levels of EYE103 in comparison with the active control, ranibizumab, in patients with diabetic macular edema (DME)

Approximately 960 participants will be entered in the study. Participants will be randomized 1:1:1 to receive low dose EYE103, high dose EYE103, or 0.5 mg ranibizumab, administered via intravitreal injection. In the first year, all 3 treatment groups will be treated every 4 weeks with either EYE103 or ranibizumab. Beginning at Year 2, the frequency of treatment for participants will shift based on a personalized treatment interval (PTI) algorithm. Throughout the 2-year study, subjects will be evaluated every 4 weeks, including measurement of ETDRS BCVA, examination by slit-lamp biomicroscopy, fundoscopy, and SD-OCT. Among other parameters, SD-OCT will be used to measure central subfield thickness (CST) in microns.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to understand the study procedures and the risks involved and provide written informed consent before the first study-related activity
* Be male or female ≥18 years of age.
* Have type 1 or type 2 diabetes mellitus and a HbA1c of ≤12%.
* Have a decrease in vision in the study eye determined by the investigator to be primarily the result of DME.

Exclusion Criteria:

* Be pregnant or breastfeeding
* History of cataract surgery and/or minimally invasive glaucoma surgery in the study eye within 90 days of Screening
* Have any treatment for complications of cataract surgery with steroids or yttrium aluminum garnet (YAG) laser capsulotomy within 90 days of Screening
* Are currently using drugs with known retinal toxicity (e.g., Hydroxychloroquine, pentosan polysulfate sodium, and amiodarone)
* If treatment-experienced for DME have a history of any of the following treatments within the noted time windows:

  * Have had prior treatment with 8 mg aflibercept (EYLEA HD) or faricimab (VABYSMO) within 120 days prior to the Screening visit in the study eye
  * Have had an IVT with other anti-VEGF treatments (ranibizumab, bevacizumab, aflibercept [2 mg], brolucizumab, pegaptanib sodium) in the study eye within 90 days of the Screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 984 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Best-Corrected Visual Acuity measured using the standardized ETDRS chart | 52 Weeks
  Change from baseline Best-Corrected Visual Acuity measured using the standardized ETDRS chart

SECONDARY OUTCOMES:
Changes in structural and visual outcomes | Duration of the study, through Week 104
  Changes in structural and visual outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Charles Miller, MD PhD, Study Director — EyeBiotech Ltd.
Locations (172):
- United States (82):
  - Scottsdale, Scottsdale, Arizona
  - Fayetteville, Arkansas, Fayetteville, Arkansas
  - Springdale, Arkansas, Springdale, Arkansas
  - Bakersfield, CA, Bakersfield, California
  - Glendale, CA, Glendale, California
  - Modesto, CA, Modesto, California
  - Mountain View, CA, Mountain View, California
  - Redlands, CA, Redlands, California
  - Sacramento, CA, Sacramento, California
  - Santa Ana, Santa Ana, California
  - Colorado Springs, CO, Colorado Springs, Colorado
  - Denver, Colorado, Denver, Colorado
  - Danbury, CT, Danbury, Connecticut
  - Manchester, CT, Manchester, Connecticut
  - Waterford,CT, Waterford, Connecticut
  - Deerfield Beach, FL, Deerfield Beach, Florida
  - Fort Lauderdale, FL, Fort Lauderdale, Florida
  - Fort Myers,FL, Fort Myers, Florida
  - Gainesville, FL, Gainesville, Florida
  - Orlando, Florida, Orlando, Florida
  - Plantation, FL, Plantation, Florida
  - Sarasota, FL, Sarasota, Florida
  - Saint Petersburg, FL, St. Petersburg, Florida
  - Tallahassee, FL, Tallahassee, Florida
  - Tampa, FL, Tampa, Florida
  - Winter Haven, FL, Winter Haven, Florida
  - Lemont, IL, Lemont, Illinois
  - Springfield, Illinois, Springfield, Illinois
  - West Des Moines, IA, West Des Moines, Iowa
  - Lenexa, Kansas, Lenexa, Kansas
  - Wichita, Kansas, Wichita, Kansas
  - Portland, Maine, Portland, Maine
  - Hagerstown, MD, Hagerstown, Maryland
  - Springfield,MA, Springfield, Massachusetts
  - Grand Rapids, Michigan, Grand Rapids, Michigan
  - Minneapolis, MN, Minneapolis, Minnesota
  - Madison, MS, Madison, Mississippi
  - Bloomfield, NJ, Bloomfield, New Jersey
  - Cherry Hill, NJ, Cherry Hill, New Jersey
  - Liverpool, NY, Liverpool, New York
  - Oceanside, NY, Oceanside, New York
  - Rochester, NY, Rochester, New York
  - Asheville, NC, Asheville, North Carolina
  - Hickory, NC, Hickory, North Carolina
  - Wake Forest, MC, Wake Forest, North Carolina
  - Winston Salem, NC, Winston-Salem, North Carolina
  - Cleveland, Ohio, Cleveland, Ohio
  - Cleveland, OH, Cleveland, Ohio
  - Youngstown, Ohio, Youngstown, Ohio
  - Edmond, OK, Edmond, Oklahoma
  - Portland, OR, Portland, Oregon
  - Springfield, Oregon, Springfield, Oregon
  - Bethlehem, PA, Bethlehem, Pennsylvania
  - Erie, PA, Erie, Pennsylvania
  - Beaufort, SC, Beaufort, South Carolina
  - Florence, SC, Florence, South Carolina
  - Ladson, SC, Ladson, South Carolina
  - West Columbia, SC, West Columbia, South Carolina
  - Germantown, TN, Germantown, Tennessee
  - Hixson, Tennessee, Hixson, Tennessee
  - Johnson City, Tennessee, Johnson City, Tennessee
  - Knoxville, TN, Knoxville, Tennessee
  - Nashville, TN, Nashville, Tennessee
  - Abilene, TX, Abilene, Texas
  - Amarillo, TX, Amarillo, Texas
  - Arlington, TX, Arlington, Texas
  - Austin, TX, Austin, Texas
  - Beaumont, TX, Beaumont, Texas
  - Bellaire, TX, Bellaire, Texas
  - Dallas, TX, Dallas, Texas
  - Fort Worth, TX, Fort Worth, Texas
  - Katy, TX, Katy, Texas
  - Plano, TX, Plano, Texas
  - Round Rock, TX, Round Rock, Texas
  - San Antonio, TX, San Antonio, Texas
  - Schertz, Texas, Schertz, Texas
  - The Woodlands, TX, The Woodlands, Texas
  - Willow Park, TX, Willow Park, Texas
  - Salt Lake City, Utah, Salt Lake City, Utah
  - Lynchburg, VA, Lynchburg, Virginia
  - Richmond, Virginia, Richmond, Virginia
  - Spokane, WA, Spokane, Washington
- Argentina (7):
  - Ciudad de Cordoba, Argentina, Córdoba, Argentina
  - Buenos Aires, Argentina, CABA, Buenos Aires
  - Caba, Buenos Aires, Argentina, Caba, Buenos Aires
  - Cordoba, Argentina, Córdoba, Córdoba Province
  - Santa Fe, Argentina, Rosario, Santa Fe Province
  - Santa Fe, Argentina, Rosario, Sante Fe
  - Buenos Aires, Argentina, CABA
- Australia (5):
  - Albury, Australia, Albury, Australia
  - Parramatta, Australia, Parramatta, Australia
  - Sydney, Australia, Sydney, Australia
  - Sydney Retina Clinic, Sydney, New South Wales
  - Sydney, Australia, Sydney, New South Wales
- Austria (4):
  - Innsbruck, Austria, Innsbruck, Austria
  - Vienna, Austria, Vienna, Vienna
  - Graz, Austria, Graz
  - Vienna, Austria, Vienna
- Colombia (5):
  - Medellin, Colombia, Medellín, Antioquia
  - Barranquilla, Colombia, Barranquilla, Atlántico
  - Medellin, Colombia, Medellín, Colombia
  - Bogota, Columbia, Bogotá, Columbia
  - Cali, Colombia, Cali, Valle del Cauca Department
- Osijek, Croatia, Osijek, Croatia
- Czechia (4):
  - Prague, Czechia, Prague, Prague
  - Mlada Boleslav, Czechia, Mladá Boleslav
  - Nachod, Czechia, Náchod
  - Prague, Czechia, Prague
- France (7):
  - Cedex, France, Dijon, Cedex
  - Lyon, France, Lyon, France
  - Paris, France, Paris, Paris
  - Creteil, France, Créteil
  - Marseille, France, Marseille
  - Paris, France, Paris
  - Saint Cyr sur Loire, France, Saint-Cyr-sur-Loire
- Germany (4):
  - Frankfurt, Germany, Frankfurt, Germany
  - Hanover, Germany, Hanover, Germany
  - Munchen, Germany, München, Germany
  - Munster, Germany, Münster, Germany
- Hungary (7):
  - Budapest, Hungary, Budapest, Budapest
  - Budapest, Hungary, Budapest, Hungary
  - Debrecen, Hungary, Debrecen, Hungary
  - Zalaegerszeg, Hungary, Zalaegerszeg, Hungary
  - Budapest, Hungry, Budapest
  - Pecs, Hungary, Pécs
  - Szeged, Hungary, Szeged
- Israel (6):
  - Rehovot, Israel, Rehovot, Israel
  - Beer Yakov, Israel, Be’er Ya‘aqov
  - Haifa, Israel, Haifa
  - Jerusalem, Israel, Jerusalem
  - Petah Tikva, Israel, Petah Tikva
  - Tel Aviv, Israel, Tel Aviv
- Italy (8):
  - Bologna, Italy, Bologna, Italy
  - Milano, Italy, Milan, Italy
  - Roma, Italy, Roma, Italy
  - Udine, Italy, Udine, Italy
  - Milano, Italy, Milan, Milano
  - Rome, Italy, Rome, Rome
  - Firenze, Italy, Florence
  - Milano, Italy, Milan
- Riga, Latvia, Riga, Rīga, Latvia
- Poland (9):
  - Gdansk, Poland, Gdansk, Gdansk
  - Bialystok, Poland, Bialystok, Poland
  - Bydgoszcz, Poland, Bydgoszcz, Poland
  - Katowice, Poland, Katowice, Poland
  - Krakow, Poland, Krakow, Poland
  - Tarnowskie Gory, Poland, Tarnowskie Góry, Poland
  - Bydgoszcz, Poland, Bydgoszcz
  - Gdansk, Poland, Gdansk
  - Olsztyn, Poland, Olsztyn
- Portugal (2):
  - Porto, Portugal, Porto, Porto District
  - Coimbra, Portugal, Coimbra
- Arecibo, PR, Arecibo, PR, Puerto Rico
- Slovakia (3):
  - Trebisov, Slovakia, Trebišov, Slovakia
  - Trencin, Slovakia, Trenčín, Slovakia
  - Zilina, Slovakia, Žilina, Slovakia
- Spain (7):
  - Barcelona, Spain, Barcelona, Barcelona
  - Sevilla, Spain, Seville, Sevilla
  - Barcelona, Spain, Barcelona, Spain
  - Santiago de Compostela, Spain, Santiago de Compostela, Spain
  - Zaragoza, Spain, Zaragoza, Spain
  - Valencia, Spain, Burjassot, Valencia
  - Barcelona, Spain, Barcelona
- Turkey (Türkiye) (2):
  - Ankara, Turkey, Ankara, Turkey
  - Balcova, Turkey, Balçova, Turkey
- United Kingdom (7):
  - London, UK, London, Middlesex
  - Bradford, United Kingdom, Bradford, United Kingdom
  - Liverpool, United Kingdom, Liverpool, United Kingdom
  - Sunderland, United Kingdom, Sunderland, United Kingdom
  - Wolverhamptom, United Kingdom, Wolverhampton, United Kingdom
  - York, United Kingdom, York, UnitedKingdom
  - Bristol, UK, Bristol

IPD SHARING:
Plan to Share IPD: No